CLINICAL TRIAL: NCT03374579
Title: Use of the Venoarterial Carbon Dioxide Gap and Arteriovenous Oxygen Content to Guide the Resuscitation in the Liver Transplant Patients
Brief Title: co2 Gap and co2/o2 Ratio in Liver Transplant Patients
Acronym: co2gap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mukhtar, Professor, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N-60-2017
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Intervention Model Description: Fluid challenge with assessment of change of co2 gap
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CO2 gap (Experimental): The patients will receive fluid bolus and observe changes in co2 gap and gap/ ratio in them.
  Interventions: Diagnostic Test: Fluid challenge

INTERVENTIONS:
Diagnostic Test: Fluid challenge — Fluid challenge and measure change in co2 gap

SUMMARY:
finding surrogate to co to trace the effect of preload challenge would make the test more applicable without the need of advanced hemodynamic monitors,suggested that co2 gap can be used to detect FR after mini fluid challenge and fluid bolts .

DETAILED DESCRIPTION:
use of carbon dioxide gap and arterio venous oxygen content to trace the effect of preload challenge by giving via a specific venous line , first 150 ml is infused over one minute, after stroke volume at one minute measure the remaining 350 ml is infused over 14 minutes at constant rate , the fluid challenge performed with albumin 5% , fluid responsiveness is an increase in stroke volume by 15% after infusion of 500ml albumin 5%.

Objectives is to investigate the ability of VA-co2 gap and gap/ ratio to predict the hemodynamic response to mini fluid challenge, and to compare the validity of VA-co2 gap and gap/ratio with svo2 for prediction of fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* patients post liver transplantation
* serum lactate >2mmol/L

Exclusion Criteria:

* age less than 18 years
* patients with fulminant liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-05-12 (Estimated); Study Completion 2018-09-12 (Estimated)

PRIMARY OUTCOMES:
co2gap | 30 minuets after fluid bolus
  Difference between arterial and venous co2 gap

SECONDARY OUTCOMES:
Stroke volume | Baseline 30 minutes after Icu admission, 1 minutes after mini fluid challenge , 30 minutes after fluid bolus
  Stroke volume assessed by cardiometry

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed m Mukhtar, professor, Principal Investigator — kasrelainy medical school,cairo university,cairo,egypt; Hassan kh Nagi, professor, Study Chair — kasrelainy medical school,cairo university,cairo,egypt
Locations (2):
- Egypt (2):
  - Cairo University Medical School, Cairo
  - Kasralainy hospital, Cairo

IPD SHARING:
Plan to Share IPD: No